CLINICAL TRIAL: NCT01283828
Title: Vaginal and Rectal Clostridial Carriage Among Women of Reproductive Age in the United States
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 7.2
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Clostridium Sordellii; Clostridium Perfringens
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal and rectal swabs
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This primary goals of this study are to: estimate the prevalence of Clostridium sordellii and Clostridium perfringens carriage in the rectum and/or vagina among women of reproductive age; estimate duration of carriage of the two clostridium species; and estimate the incidence of carriage at 2 weeks after a negative test.

DETAILED DESCRIPTION:
Since 2000, clostridial pelvic infections have claimed the lives of at least 17 young, previously healthy women. The majority of infections detected by molecular methods were among women testing positive for Clostridium sordellii only; in 5 cases, deaths were due to Clostridium perfringens only; and in 3 cases, the women were positive for both. These deaths occurred among both non-pregnant and recently pregnant women. Clostridium has been isolated from the vagina in 4-18% of normal, health non-pregnant women, with Clostridium perfringens the most common isolate. Most studies do not differentiate the small percentage of other clostridia present in the vaginal microenvironment. The vaginal carriage rate for Clostridium sordellii remains unknown, but is probably very low, less than 1%.

The correlates of clostridial carriage are unknown, and data on the etiology and lethality of clostridial infection among women of reproductive age are insufficient to guide possible courses of safe and effective prevention. In women infected with strains of Clostridium perfringens and Clostridium sordellii that produce the lethal toxin, it is not clear whether there is an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Between ages 18 and 45

Exclusion Criteria:

-Seeking emergency or oncological care

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Approximately 5,000 women aged 18 to 45 years in the United States will be enrolled in the study. Women will be recruited from approximately 25 clinics and solo or group practices providing maternity care (pre- and post-natal), abortion, STI prevention & treatment, family planning, and student health services. All women will be recruited, excluding women seeking emergency or oncological care.
Sampling Method: Non-Probability Sample
Enrollment: 4977 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of C sordellii or C perfringens carriage in the rectum/vagina | 2 years

SECONDARY OUTCOMES:
Duration of carriage of C sordellii or C perfringens | 2 years
Incidence of C. sordelli or C. perfringens carriage at 2 weeks after a negative test | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, M.D., M.P.H., Principal Investigator — Gynuity Health Projects
Locations (18):
- United States (18):
  - Montgomery Women's Health Associates, Montgomery, Alabama
  - University of Arizona, Tucson, Arizona
  - Planned Parenthood of the Rocky Mountains, Boulder, Colorado
  - UC Denver- Comprehensive Women's Health Center, Denver, Colorado
  - Feminist Women's Center, Atlanta, Georgia
  - Family Planning Associates Medical Group, Chicago, Illinois
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - Women's Health Research Center, Plainsboro, New Jersey
  - Mt Sinai Medical Center, New York, New York
  - Red River Women's Clinic, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Downtown Gynecology, Portland, Oregon
  - Downtown Women's Center, Portland, Oregon
  - Philadelphia Women's Center, Philadelphia, Pennsylvania
  - Whole Women's Health of Fort Worth, Fort Worth, Texas
  - Dr Barry Troyan, Houston, Texas
  - Dairy Ashford Family Practice, Houston, Texas
  - Cedar River Clinic, Seattle, Washington

REFERENCES:
- [Derived] Chong E, Winikoff B, Charles D, Agnew K, Prentice JL, Limbago BM, Platais I, Louie K, Jones HE, Shannon C; NCT01283828 Study Team. Vaginal and Rectal Clostridium sordellii and Clostridium perfringens Presence Among Women in the United States. Obstet Gynecol. 2016 Feb;127(2):360-8. doi: 10.1097/AOG.0000000000001239. PMID 26942366